CLINICAL TRIAL: NCT07111286
Title: Impact of Motor Imagery in the Functional Rehabilitation of Patients With Chronic Low Back Pain: a Randomised Controlled Trial
Acronym: MIRACLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GUEUGNON CRBFC 2023
Record Dates: First submitted 2025-07-31; First posted 2025-08-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Common Non-specific Low Back Pain
MeSH Terms: interventions — Restraint, Physical; Drug Tolerance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with motor imagery (Experimental)
  Interventions: Other: Assessment; Other: Motor imagery task sessions; Other: Assessment of satisfaction and tolerance
- Control (Active Comparator)
  Interventions: Other: Assessment; Other: Cognitive task sessions

INTERVENTIONS:
Other: Assessment — Before and after the programme :
  * Self-questionnaires: assessment of pain (visual analogue scale), functional disability (Oswestry), kinesiophobia (Tampa scale of Kinesiophobia), mood (Hospital Anxiety Depression Scale), quality of life (SF12), level of physical activity (Simple Physical Activity Questionnaire), and level of motor imagery (Kinesthesic and Visual Imagery Questionnaire-10)
  * Functional tests: Sorensen test, Shirado test, Time Up and Go test (TUG), 6-minute walk test, 200-metre fast walk test, measurement of maximum isometric strength of back extensors/flexors, 3D analysis of locomotion, posture and trunk flexion.
  * Evaluation of excitability and inhibition mechanisms within the primary motor cortex at rest and during motor imagery using single and double pulse TMS. Excitability between the brain and the erector spinae muscles and inhibition of the primary motor cortex will be measured at rest and during imagery of back flexion and extension movements
Other: Motor imagery task sessions — 3 sessions of 30 minutes per week
  Arms: Group with motor imagery
Other: Cognitive task sessions — 3 sessions of 30 minutes per week
  Arms: Control
Other: Assessment of satisfaction and tolerance — During the final assessment, which will take place after the programme. Satisfaction and tolerance will be assessed using a visual analogue scale.
  Arms: Group with motor imagery

SUMMARY:
Non-specific low back pain (NSLBP) is a very common condition and one of the leading causes of disability worldwide. It has a significant impact on quality of life, with functional, locomotor and psychological repercussions, and is often associated with kinesiophobia (excessive fear of movement due to apprehension related to pain or injury). For the most severe cases, multidisciplinary rehabilitation programmes are recommended. The objectives are, on the one hand, to offer reconditioning to exercise and, on the other hand, to educate, raise awareness about physical activity and help combat fears in order to reduce symptoms, improve quality of life and re-engage in daily and professional activities. However, these programmes are not entirely effective, and many of you still live with chronic lower back pain.

To improve the management of lower back pain, it is important to understand how the body functions with this condition, particularly when there is chronic pain. It has been shown that people suffering from lower back pain often have difficulty controlling their movements. This means that their brain is less able to prepare certain movements. One method that can help improve movement preparation and control is motor imagery (MI). This involves imagining a movement without physically performing it. This technique activates the same areas of the brain as when the movement is performed. This is why it can be beneficial and help improve treatment.

This research will evaluate the effectiveness of an innovative rehabilitation programme incorporating motor imagery (MI) in patients with chronic low back pain. MI could improve motor skills at the end of rehabilitation as well as quality of life. Conversely, the inability to perform certain movements, kinesiophobia and pain could be reduced.

Each participant will follow the REAGIR multimodal rehabilitation programme at the Dijon Bourgogne University Hospital (7 hours of rehabilitation per day, 5 days per week for 3 weeks, consisting of activities such as: personalised whole-body exercises (aerobic) on ergometers; resistance training, balneotherapy, therapeutic education, individual and group motivational interviews, nutritional advice, relaxation sessions and psychology sessions). By participating in this study, patients will benefit from this programme as well as 30-minute motor imagery sessions, the content of which will depend on the experimental group to which they are assigned after randomisation.

Participation will also include a visit before the start and after the end of the programme in order to carry out various assessments.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Person who has given their verbal consent
* Suffering from chronic non-specific low back pain that has been ongoing for more than 6 months
* Eligible for a multimodal rehabilitation programme according to the investigating physician

Exclusion Criteria:

* Persons not affiliated with or not covered by a social security scheme
* Patients subject to legal protection measures (guardianship, curatorship)
* Patients subject to judicial protection measures
* Pregnant women, women in labour or breastfeeding women
* Adults who are incapacitated or unable to give their consent
* Patients with a history of repeated falls
* Scheduled lumbar spine surgery in the coming year
* Associated conditions other than spinal conditions (orthopaedic, neurological, vascular, cardiac, etc.) that could significantly impair mobility
* Radicular involvement (sciatica or cruralgia) with motor deficit < 3 in the lower limbs
* Impaired comprehension skills making self-assessment impossible
* Patients with poorly controlled epilepsy
* Individuals who are not fluent in English
* Patients who have already completed a multimodal rehabilitation programme in a specialised centre

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Duration in seconds during the functional endurance test of the trunk extensors (Sorensen test) | At baseline (Month 1) and Month 3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France